CLINICAL TRIAL: NCT01997567
Title: Are Preemptive Femoral and Lateral Femoral Cutaneous Nerve Blocks Given Immediately Prior to Hip Arthroscopy(THA) Effective for Acute Postoperative Pain Management?
Brief Title: Preemptive Femoral & Lateral Femoral Cutaneous Nerve Blocks for THA Acute Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Subject recruitment is too difficult and we foresee that this will not improve
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Sandeep Amin, MD, Assistant Professor, Attending Anesthesiologist, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Hip-Scope-Block
Record Dates: First submitted 2013-06-13; First posted 2013-11-28 (Estimated); Results first posted 2016-06-17 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Internal Derangement of Hip; Acetabular Labrum Tear
Keywords: Hip Arthroscopy; Regional Anesthesia; Peripheral Nerve block
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grp 1 Ropivacaine Block (Active Comparator): Group 1 consented subjects will receive for their hip arthroscopy procedures general anesthesia (sevoflurane) with single femoral and lateral femoral cutaneous nerve blocks under ultrasound guidance, with 20 ml solution for the femoral block and 10 ml for lateral femoral cutaneous block, for a total of 30 ml solution of ropivacaine 0.5% with epinephrine 1:200,000 (150mcg) as a tracer for intravascular injection (total 30 ml)
  Interventions: Drug: Ropivacaine
- Grp 2 Placebo Block (Placebo Comparator): Group 2 consented subjects will receive for their hip arthroscopy procedures general anesthesia (sevoflurane) with single femoral and lateral femoral cutaneous nerve blocks under ultrasound guidance, with 20 ml solution for the femoral block and 10 ml for lateral femoral cutaneous block, for a total of 30 ml solution of saline with epinephrine 1:200,000 (150 mcg) (total 30 ml)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ropivacaine — Subjects will receive for their hip arthroscopy procedures general anesthesia (sevoflurane) with single femoral and lateral femoral cutaneous nerve blocks under ultrasound guidance, with 20 ml solution for the femoral block and 10 ml for lateral femoral cutaneous block, for a total of 30 ml solution of ropivacaine 0.5% with epinephrine 1:200,000 (150mcg) as a tracer for intravascular injection (total 30 ml)
  Arms: Grp 1 Ropivacaine Block
Drug: Placebo — Group 2 consented subjects will receive for their hip arthroscopy procedures general anesthesia (sevoflurane) with single femoral and lateral femoral cutaneous nerve blocks under ultrasound guidance, with 20 ml solution for the femoral block and 10 ml for lateral femoral cutaneous block, for a total of 30 ml solution of saline with epinephrine 1:200,000 (150 mcg) (total 30 ml)
  Arms: Grp 2 Placebo Block

SUMMARY:
The goal of the study is to evaluate via a prospective, blinded, randomized clinical trial, whether ultrasound-guided single femoral and lateral femoral cutaneous nerve blocks with ropivacaine 0.5% with epinephrine (1:200,000) as a tracer for intravascular injection (total 30 ml) vs. saline with epinephrine (1:200,000) (total 30 ml), given just prior to same day elective hip arthroscopy, is effective in reducing acute postoperative pain (NRS scores), postoperative opiate consumption, and time to discharge from the postanesthesia care unit. Differences between groups with respect to postoperative quality of life and functional scores will also be evaluated.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether ultrasound (using sound waves to produce an image)-guided regional anesthesia (local numbing medicine) to the hip area given in addition to general anesthesia just prior to same day elective hip arthroscopy, is effective in reducing acute postoperative pain, and time to discharge from the post anesthesia care unit. In addition, the study aims to examine whether this regional anesthesia medication has any effect on the study subjects' use of pain medication both during and after the procedure, return to function, and quality of life in the 6 month period after the surgical procedure. Although hip arthroscopy is a routine procedure, the best method for pain control is not well established, and is the purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* >18 year old,
* ASA physical status classification system score (ASA) <=3
* due to undergo elective unilateral hip arthroscopy by one surgeon Dr. Nho (Co-Principal Investigator)

Exclusion Criteria:

* ASA physical status classification system score) (ASA) >3
* history of opioid dependence or abuse
* current chronic analgesic therapy (daily use =>20 mg oxycodone-equivalent opioid use within 2 weeks before surgery and duration of use >=4 weeks)
* allergy to study medications (fentanyl and ropivicaine)
* any neuromuscular deficit of the ipsilateral femoral nerve or quadriceps femoris muscle (including diabetic peripheral neuropathy)
* diagnosis of hypertension and/or current treatment for hypertension
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Amin, M.D., Principal Investigator — Rush University Medical Center; Shane Nho, M.D., M.S., Principal Investigator — Rush University Medical Center
Locations (1):
- Rush Oak Park Hospital, Oak Park, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No data to Share

REFERENCES:
- [Background] YaDeau JT, Tedore T, Goytizolo EA, Kim DH, Green DS, Westrick A, Fan R, Rade MC, Ranawat AS, Coleman SH, Kelly BT. Lumbar plexus blockade reduces pain after hip arthroscopy: a prospective randomized controlled trial. Anesth Analg. 2012 Oct;115(4):968-72. doi: 10.1213/ANE.0b013e318265bacd. Epub 2012 Jul 19. PMID 22822195
- [Background] Ward JP, Albert DB, Altman R, Goldstein RY, Cuff G, Youm T. Are femoral nerve blocks effective for early postoperative pain management after hip arthroscopy? Arthroscopy. 2012 Aug;28(8):1064-9. doi: 10.1016/j.arthro.2012.01.003. Epub 2012 Apr 11. PMID 22498045
- [Background] Lee EM, Murphy KP, Ben-David B. Postoperative analgesia for hip arthroscopy: combined L1 and L2 paravertebral blocks. J Clin Anesth. 2008 Sep;20(6):462-5. doi: 10.1016/j.jclinane.2008.04.012. PMID 18929290
- [Background] Good RP, Snedden MH, Schieber FC, Polachek A. Effects of a preoperative femoral nerve block on pain management and rehabilitation after total knee arthroplasty. Am J Orthop (Belle Mead NJ). 2007 Oct;36(10):554-7. PMID 18033568
- [Background] Aprato A, Jayasekera N, Villar R. Timing in hip arthroscopy: does surgical timing change clinical results? Int Orthop. 2012 Nov;36(11):2231-4. doi: 10.1007/s00264-012-1655-x. Epub 2012 Sep 11. PMID 22965491

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Grp 1 Ropivacaine Block | Grp 2 Placebo Block
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was closed due to enrollment issues and data were not collected or analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Grp 1 Ropivacaine Block | Grp 2 Placebo Block | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Pain Numerical Rating Scale Score (NRS 0-10)
Description: The primary outcome measure will be pain scores at rest (NRS 0-10). Those scores will be documented at initial visit prior to surgery, and at postoperative office visits at 3 weeks, 3 months and 6 months post-procedure.
Time Frame: Preoperative 2-8 wks
Population: Study was closed due to enrollment issues and data were not collected or analyzed.
Arm/Group | Grp 1 Ropivacaine Block | Grp 2 Placebo Block
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Pain Numerical Rating Scale Score (NRS 0-10)
Description: The primary outcome measure will be pain scores at rest (NRS 0-10). Those scores will be documented at initial visit prior to surgery, and at postoperative office visits at 3 weeks, 3 months and 6 months post-procedure.
  Study was closed due to enrollment issues and data were not collected or analized.
Time Frame: 3 wks postoperative
Population: Study was closed due to enrollment issues and data were not collected or analized.
Arm/Group | Grp 1 Ropivacaine Block | Grp 2 Placebo Block
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Pain Numerical Rating Scale Score (NRS 0-10)
Description: as for outcome 1
Time Frame: 3 months postoperative
Population: Study was closed due to enrollment issues and data were not collected or analyzed.
Arm/Group | Grp 1 Ropivacaine Block | Grp 2 Placebo Block
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Pain Numerical Rating Scale Score (NRS 0-10)
Description: as for outcome 1
Time Frame: 6 months postoperative
Population: Study was closed due to enrollment issues and data were not collected or analyzed.
Arm/Group | Grp 1 Ropivacaine Block | Grp 2 Placebo Block
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Veterans Research and Development (RAND) 12 Item Health Survey (VR-12) Scores
Description: Preoperative VR-12 scores will be compared with the VR-12 scores obtained at the 3 mo and 6 mo postoperative visits.
Time Frame: Preoperative 2-8 wks
Population: Study was closed due to enrollment issues and data were not collected or analyzed.
Arm/Group | Grp 1 Ropivacaine Block | Grp 2 Placebo Block
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Veterans RAND 12 Item Health Survey (VR-12) Scores
Description: Preoperative VR-12 scores will be compared with the VR-12 scores obtained at the 3 mo and 6 mo postoperative visits.
Time Frame: 3 months postoperative
Population: Study was closed due to enrollment issues and data were not collected or analyzed.
Arm/Group | Grp 1 Ropivacaine Block | Grp 2 Placebo Block
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Veterans RAND 12 Item Health Survey (VR-12) Scores
Description: Preoperative VR-12 scores will be compared with the VR-12 scores obtained at the 3 mo and 6 mo postoperative visits.
Time Frame: 6 months postoperative
Population: Study was closed due to enrollment issues and data were not collected or analyzed.
Arm/Group | Grp 1 Ropivacaine Block | Grp 2 Placebo Block
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: None. Study closed and data not collected
Arm/Group | Grp 1 Ropivacaine Block | Grp 2 Placebo Block
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes